CLINICAL TRIAL: NCT00264225
Title: A Randomized, Double-Blind, Comparative Parallel Group Study of Analgesic Effectiveness and Safety of Three Different Doses of Lamaline® New Formulation vs Dafalgan® Codeine, After 10 Days Administration in Subjects With Painful Gonarthrosis.
Brief Title: Analgesic Effectiveness of Three Different Doses of a New Formulation of Lamaline in a Model of Painful Knee (Gonarthrosis)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S118.3.005; 2005-003757-27
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2008-02

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis, pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

INTERVENTIONS:
Drug: Lamaline® , 3 different doses, Dafalgan codeine

SUMMARY:
This study aims to assess the analgesic effectiveness and safety of three different doses of a new formulation of Lamaline® versus Dafalgan® Codeine after 10 days administration in subjects with painful gonarthrosis

ELIGIBILITY:
Inclusion Criteria:

* History of knee (unilateral or bilateral) osteoarthritis for at least 6 months
* Pain intensity assessed by Visual Analogue Scale ≥ 40 mm
* Partial functional disability assessed by Lequesne index ≥4 and < than 12

Exclusion Criteria:

* Patient unable to interrupt his/her NSAIDs to participate in the clinical study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (171):
- France (171):
  - Site 2, Albi
  - Site 3, Andernos-les-Bains
  - Site 101, Angers
  - Site 103, Angers
  - Site 105, Angers
  - Site 106, Angers
  - Site 107, Angers
  - Site 108, Angers
  - Site 109, Angers
  - Site 110, Angers
  - Site 117, Angers
  - Site 121, Angers
  - Site 123, Angers
  - Site 124, Angers
  - Site 129, Angers
  - Site 134, Angers
  - Site 138, Angers
  - Site 140, Angers
  - Site 453, Angers
  - Site 496, Angers
  - Site 498, Angers
  - Site 215, Anzin
  - Site 451, Avrillé
  - Site 131, Bagneux
  - Site 315, Bandol
  - Site 4, Bassens
  - Site 115, Beaucouzé
  - Site 502, Beaumont-sur-Lèze
  - Site 449, Beaupréau
  - Site 213, Bersée
  - Site 119, Bécon-les-Granits
  - Site 135, Bécon-les-Granits
  - Site 136, Bécon-les-Granits
  - Site 506, Bérat
  - Site 50, Béziers
  - Site 55, Béziers
  - Site 5, Bobigny
  - Site 6, Bordeaux
  - Site 122, Briollay
  - Site 7, Brive-la-Gaillarde
  - Site 8, Carpentras
  - Site 76, Châlons-en-Champagne
  - Site 9, Châlons-en-Champagne
  - Site 432, Château-Gontier
  - Site 433, Château-Gontier
  - Site 48, Châtenay-Malabry
  - Site 114, Chemillé-Melay
  - Site 462, Cherbourg
  - Site 10, Clamart
  - Site 11, Clermont-Ferrand
  - Site 12, Clermont-Ferrand
  - Site 13, Clermont-Ferrand
  - Site 14, Colmar
  - Site 78, Colmar
  - Site 219, Croix
  - Site 15, Dijon
  - Site 16, Dinan
  - Site 17, Dinard
  - Site 47, Dinard
  - Site 507, Eaunes
  - Site 120, Écouflant
  - Site 18, Évreux
  - Site 19, Évreux
  - Site 46, Évreux
  - Site 102, Fenioux
  - Site 20, Fontenay Malabry
  - Site 24, L'Union
  - Site 306, La Garde
  - Site 207, La Riche
  - Site 209, La Riche
  - Site 423, La Rochelle
  - Site 318, La Seyne-sur-Mer
  - Site 319, La Seyne-sur-Mer
  - Site 320, La Seyne-sur-Mer
  - Site 321, La Seyne-sur-Mer
  - Site 454, Laval
  - Site 458, Laval
  - Site 459, Laval
  - Site 460, Laval
  - Site 461, Laval
  - Site 224, Le Pradet
  - Site 225, Le Pradet
  - Site 118, Les Ponts-de-Cé
  - Site 137, Les Ponts-de-Cé
  - Site 21, Levallois-Perret
  - Site 22, Libourne
  - Site 23, Limoges
  - Site 49, Lyon
  - Site 53, Lyon
  - Site 58, Lyon
  - Site 59, Lyon
  - Site 64, Lyon
  - Site 25, Marseille
  - Site 26, Marseille
  - Site 27, Marseille
  - Site 28, Marseille
  - Site 77, Marseille
  - Site 29, Mérignac
  - Site 70, Millau
  - Site 56, Montpellier
  - Site 60, Montpellier
  - Site 62, Montpellier
  - Site 65, Montpellier
  - Site 68, Montpellier
  - Site 139, Montreuil-Bellay
  - Site 133, Montrevault
  - Site 30, Montrouge
  - Site 51, Nice
  - Site 54, Nice
  - Site 57, Nice
  - Site 61, Nice
  - Site 71, Nice
  - Site 74, Nice
  - Site 63, Nîmes
  - Site 67, Nîmes
  - Site 69, Nîmes
  - Site 73, Nîmes
  - Site 130, Noyant
  - Site 128, Parçay-les-Pins
  - Site 31, Paris
  - Site 32, Paris
  - Site 66, Perpignan
  - Site 33, Pont-de-l'Arche
  - Site 34, Rennes
  - Site 52, Rennes
  - Site 75, Rodez
  - Site 35, Roquebrune-Cap-Martin
  - Site 36, Rosny-sous-Bois
  - Site 202, Saint-Avertin
  - Site 208, Saint-Avertin
  - Site 457, Saint-Berthevin
  - Site 489, Saint-Brice-Courcelles
  - Site 313, Saint-Mandrier-sur-Mer
  - Site 113, Segré
  - Site 413, Seysses
  - Site 414, Seysses
  - Site 494, Seysses
  - Site 495, Seysses
  - Site 314, Six-Fours-les-Plages
  - Site 37, Six-Fours-les-Plages
  - Site 38, Six-Fours-les-Plages
  - Site 39, Strasbourg
  - Site 40, Strasbourg
  - Site 79, Strasbourg
  - Site 132, Thouars
  - Site 104, Tiercé
  - Site 126, Tiercé
  - Site 221, Toulon
  - Site 228, Toulon
  - Site 301, Toulon
  - Site 302, Toulon
  - Site 316, Toulon
  - Site 41, Toulouse
  - Site 42, Toulouse
  - Site 43, Toulouse
  - Site 44, Toulouse
  - Site 45, Toulouse
  - Site 503, Toulouse
  - Site 511, Toulouse
  - Site 201, Tours
  - Site 204, Tours
  - Site 401, Tours
  - Site 402, Tours
  - Site 405, Tours
  - Site 410, Tours
  - Site 112, Trélazé
  - Site 116, Trélazé
  - Site 72, Vernet-les-Bains
  - Site 488, Verzy
  - Site 125, Vihiers
  - Site 127, Villebernier